CLINICAL TRIAL: NCT02760849
Title: WISP (Women Choosing Surgical Prevention)
Brief Title: Surgery in Preventing Ovarian Cancer in Patients With Genetic Mutations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0814; NCI-2016-00778 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0814 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Deleterious BARD1 Gene Mutation; Deleterious BRCA1 Gene Mutation; Deleterious BRCA2 Gene Mutation; Deleterious BRIP1 Gene Mutation; Deleterious EPCAM Gene Mutation; Deleterious MLH1 Gene Mutation; Deleterious MSH2 Gene Mutation; Deleterious MSH6 Gene Mutation; Deleterious PALB2 Gene Mutation; Deleterious PMS2 Gene Mutation; Deleterious RAD51C Gene Mutation; Deleterious RAD51D Gene Mutation; Hereditary Breast and Ovarian Cancer Syndrome; Premenopausal
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Ovariectomy; Salpingectomy; Salpingo-oophorectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ISDO) (Experimental): Patients undergo ISDO.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Oophorectomy; Other: Quality-of-Life Assessment; Procedure: Salpingectomy
- Arm II (RRSO) (Active Comparator): Patients undergo RRSO.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Procedure: Salpingo-Oophorectomy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Oophorectomy — Undergo ISDO
  Other Names: Female Castration; Ovariectomy
  Arms: Arm I (ISDO)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Salpingectomy — Undergo ISDO
  Other Names: Tubal Excision
  Arms: Arm I (ISDO)
Procedure: Salpingo-Oophorectomy — Undergo RRSO
  Arms: Arm II (RRSO)

SUMMARY:
This phase II trial studies how well surgery works in preventing ovarian cancer in patients with genetic mutations at risk of ovarian cancer. Risk reducing salpingo oophorectomy (RRSO) is surgery to remove the fallopian tubes and ovaries at the same time. Interval salpingectomy with delayed oophorectomy (ISDO) is surgery to remove the fallopian tubes. It is not known whether ISDO works better than RRSO at lowering risk of ovarian cancer and improving the sexual function and psychosocial well-being in patients with genetic mutation.

DETAILED DESCRIPTION:
Primary Objectives:

1. To examine changes in female sexual function with the strategy of interval salpingectomy and delayed oophorectomy (ISDO) compared to the strategy of risk-reducing salpingo-oophorectomy (RRSO) for patients who carry genetic mutations that predispose them to ovarian cancer.

Secondary Objectives:

1. To estimate the onset and severity of menopausal symptoms with ISDO compared to RRSO.
2. To estimate quality of life with ISDO compared to RRSO.
3. To examine participants' satisfaction level and cancer worry level with their choice of prophylactic procedures.
4. To estimate the impact of ISDO compared to RRSO on mental health, including depression, anxiety, and sleep quality.
5. To determine the compliance with delayed oophorectomy within the ISDO arm.
6. To estimate the number of fallopian tube, ovarian, primary peritoneal malignancies and other malignancies over the course of the study.
7. To identify common themes regarding influential factors in the decision to undergo risk reducing surgery in premenopausal women at genetic high-risk for ovarian can

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients undergo ISDO.

ARM II: Patients undergo RRSO.

After completion of study treatment, patients are followed up at 1 and 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women must be ≥ 30 and ≤ 50 years of age.
2. Premenopausal women with a documented deleterious mutation in one of the following ovarian cancer genes: BRCA1, BRCA2, BRIP1, PALB2, RAD51C, RAD51D, BARD1, MSH2, MSH6, MLH1, PMS2, or EPCAM. Menopause is defined as ≥ 12 months of amenorrhea. However, for those patients with ≥ 12 months of amenorrhea who may be pre-menopausal, levels of FSH, LH, and estradiol in the pre-menopausal range will be acceptable.
3. Willing to undergo two surgical procedures (if chooses the ISDO arm).
4. Presence of at least 1 fallopian tube and 1 ovary. Prior unilateral salpingectomy is allowed; prior bilateral salpingectomy is not allowed
5. Patients who have undergone a prior tubal ligation will be eligible.
6. Participants may have a personal history of non-ovarian malignancy, but must:

   1. Be without evidence of disease at enrollment
   2. Remain premenopausal
   3. Have completed treatment (including surgery, chemotherapy, radiotherapy or hormonal therapy) > 3 months prior to enrollment (other than non-melanoma skin cancer)
7. Willingness to return to the enrolling site for the study surgical procedures, including pre-operative and post-operative care.

   Patients in the ISDO arm must be willing to return to the enrolling site for yearly ovarian cancer assessment.
8. Patients must understand that they will be permanently sterilized

Exclusion Criteria:

1. Women with a personal history of ovarian, fallopian tube, or primary peritoneal cancer.
2. Current treatment with Tamoxifen or Aromatase Inhibitors.
3. Medical comorbidities making surgery unsafe as determined by the patient's surgeon.
4. Women who are pregnant or post-partum (within 3 months of delivery).

   * Patients are deemed not pregnant by virtue of urine pregnancy test (UPT), transvaginal ultrasound, beta HCG, or best judgment of the investigator. Pregnancy testing is not required per protocol to determine study eligibility.
   * Women who become pregnant on the ISDO arm via reproductive technology can remain on study. However, data collection will be suspended during pregnancy and 3 months post-partum.
5. Women with elevated levels of CA125 (>50) or transvaginal ultrasound suggesting cancer, unless findings are consistent with endometriosis. CA125 and transvaginal ultrasounds must be the most recent, but no older than 1 year from the date of enrollment.
6. Inability to provide informed consent.
7. Inability to read or speak English.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2041-05-31 (Estimated); Study Completion 2041-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent of women with clinically meaningful change in the Female Sexual Function Index (FSFI) score | From baseline to 6 months
  Will be calculated using the Cochran-Mantel-Haenszel test stratified by age, with 5-year age groups. We will use propensity score methods to account for potential differences between interval salpingectomy with delayed oophorectomy (ISDO) and risk-reducing bilateral salpingectomy with oophorectomy (RRSO) arms with respect to age, baseline survey scores, and other potential confounders, and we will use the propensity scores as inverse weights in logistic regression to model the logit of the probability of having a clinically meaningful change in FSFI score from baseline to 6 months as our primary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Roni N Wilke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: WISP University of Texas M D Anderson Cancer Center — http://www.mdanderson.org